CLINICAL TRIAL: NCT01406366
Title: Evaluation of a Bright Futures Oral Health Intervention for Pediatric Residents
Brief Title: Evaluation of a Bright Futures Oral Health Intervention
Acronym: BFOH
Status: Completed | Type: Observational
Sponsor: Continuity Research Network (Network)
Responsible Party: Henry Bernstein DO, Principal Investigator, CORNET, Academic Pediatric Association
Other Study IDs: R40MC05267-01-00; R40MC05267-01-00 (Other Grant/Funding Number: MCHB)
Record Dates: First submitted 2011-07-29; First posted 2011-08-01 (Estimated); Last update posted 2011-08-01 (Estimated); Status verified 2010-08

CONDITIONS: Health Knowledge, Attitudes, Practice
Keywords: Pediatric oral health; Bright Futures; Health promotion
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1: Group 1: 16 programs / 148 residents
  Interventions: Behavioral: Group 1: Bright Futures Oral Health Curriculum
- Group 2: Group 2: 16 programs / 142 residents
  Interventions: Behavioral: Group 2: Iron Deficiency Training Module

INTERVENTIONS:
Behavioral: Group 1: Bright Futures Oral Health Curriculum — Residents who are randomized to Group 1 will receive a resident curriculum that exposes them to Bright Futures concepts of health promotion, including partnership building, communication and oral health. Group 1 residents will complete 7 modules, 3 on Bright Futures concepts (health, partnership building and communication), and 4 on oral health promotion. These modules have been developed in collaboration with the Pediatrics in Practice workgroup and the Open Wide modules endorsed by the American Academy of Pediatrics and the Maternal and Child Health Bureau. The oral health modules address dental caries development and prevention, importance of identifying maternal oral health status, duration of bottle-feeding or breastfeeding and discouraging both during sleep.
  Groups: Group 1
Behavioral: Group 2: Iron Deficiency Training Module — Our study team opted to include a single 1-hour educational module addressing the identification and prevention of iron deficiency created by the AAP on Pedialink® to the active control group. This educational module addresses screening for and assessing risk for iron deficiency.
  Groups: Group 2

SUMMARY:
Pediatricians serve an important role in promoting health in families. Bright Futures offers a child and family-centered approach to health promotion in incorporating partnership and communication skills of providers. Two areas of importance are in promotion of oral health and prevention of iron deficiency. We plan to study implementing educational curriculum to pediatric residents through a randomized controlled trial. Randomization will be done through assignment at the level of pediatric training program. Residents randomized to Group 1 will receive education about Bright Futures partnership and communication skills with oral health as the main health promotion topic. Group 2 will receive educational curriculum pertaining to the topic of iron deficiency prevention. While pediatricians are positioned perfectly to partner and effectively communicate with families on these two issues, there are gaps in pediatric education addressing these topics. The CORNET continuity practices of the Ambulatory Pediatric Association provide a venue through which multiple residency programs that educate pediatric residents and whose residents provide medical care to underserved children can participate. The research hypotheses include:

1. Residents in Group 1 will have greater confidence, knowledge and competence in partnership building and communication with families
2. Residents in Group 1 will have greater knowledge and competence in discussing oral health promotion
3. Residents in Group 2 will have greater knowledge and competence in discussing iron deficiency prevention
4. Parent-child dyads in Group 1 will be more likely to have established a dental home
5. Parent-child dyads in Group 1 will be more likely to be satisfied with their healthcare encounter.

Pediatric practices provide fertile ground for the provision of health promotion on oral health and iron deficiency prevention. However, evidence for the effectiveness of primary care clinician interventions of screening, referral and counseling to prevent dental caries is lacking [14]. The National Survey of America's Families [15] found 47% of children did not receive the recommended number of dental visits, with the youngest ones being least likely to receive any dental care.

Although 90% of pediatricians agreed they had important roles in identifying and counseling patients on prevention of caries, half stated they had received no previous training during medical school or residency and their knowledge of basic oral health topics was limited [13]. These studies highlight that pediatricians play important roles in oral health and are capable of being trained to complete oral screening exams, but more education and guidance is needed.

Iron deficiency is the most common childhood nutritional deficiency in the United States. Recent prevalence data have determined that 7-30% of children in the United States aged 1-2 years have iron deficiency and 3-10% have iron deficiency anemia [17, 18]. Specific goals in Health People 2010 include a reduction of iron deficiency to 5% in children less than 3 years of age.

DETAILED DESCRIPTION:
Although health professionals must be equipped to promote healthy lifestyles and serve as resources for the public's health information, many gaps in the education and training of residents exist. Health professional students readily admit to deficiencies in their training (i.e. lack of learning principles of prevention, health promotion, behavior change and risk reduction), yet, curricular changes have been slow [1,2]. A 1997 AAMC Medical School Graduation Questionnaire revealed that almost one quarter of graduates felt instruction time devoted to health promotion and disease prevention was inadequate [3, 4, 5, 6]. Mandates for competency-based, post-graduate training by the ACGME Outcomes Project and competency expectations by the AAMC Medical Schools Objectives Project (MSOP) require all residency programs and medical schools to develop innovative approaches to teaching clinical skills.

We believe the resident continuity experience is the perfect venue to implement and practice clinical guidelines and Bright Futures concepts. Past studies have documented that residents in academic, hospital-based sites, similar to those in CORNET, experience the most continuity and longitudinal relationships with their patients [7, 8, 9]. Longitudinal learning is a basic tenet of successful interventions and is easily accomplished during resident continuity practice. Pediatrics in Practice provides key resources for enhancing knowledge in family-centered oral health promotion and responding to the present gaps in medical education and training. Both residents and pediatricians in practice have limited knowledge of Bright Futures and its tenets. Bright Futures: Guidelines for Health Supervision of Infants, Children, and Adolescents represents the framework of providing contextual care to children that fosters partnerships among families, health professionals, and communities and increases knowledge about health education and prevention [10, 11, 12]. Although more competency-based curricula are being designed to promote skills and knowledge in health promotion and preventive services, there has been very little research into their efficacy in trainees.

ELIGIBILITY:
Inclusion Criteria:

* Residents

  1. Pediatric categorical residents
  2. PL-1 or PL-2 level
* Parents/Patients

  1. Parents/legal guardian of children 12- 35 months of age
  2. Legal guardian present at visit
  3. Primary care provider is pediatric resident seeing patient at that visit
  4. Child presents for health maintenance visit
  5. English speaking

Ages: 12 Months to 35 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Pediatric categorical residents in continuity clinics associated with CORNET practices that volunteer to participate will be asked to participate in the study. Resident inclusion criteria will include pediatric residents in their 1st or 2nd year of categorical training. Parent-child dyad inclusion criteria include children between 12-35 months of age, accompanied by a legal guardian, who presents for a scheduled health maintenance visit with their primary care provider who is a pediatric resident. Families must have a means by which to be contacted (i.e., telephone, cell phone, or beeper number) for follow-up. At least 2 numbers for communication will need to be solicited.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2005-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry H Bernstein, DO, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth Hitchcock Medical Center, Hanover, New Hampshire, United States

REFERENCES:
- See also: A Bright-Futures based website supporting faculty in health promotion — http://www.pediatricsinpractice.org